CLINICAL TRIAL: NCT00993603
Title: The Effect of an 8-month Intensive Lifestyle Intervention on Hormonal Factors Regulating Food Intake in Obese, Non-diabetic Adults With a Family History of Diabetes.
Brief Title: Lifestyle Intervention in Obese Non-diabetic Adults With a Family History of Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Non-DM Lifestyle.; REC reference: 09/H0504/61
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Lifestyle; Diabetes Mellitus; prevention/onset delay.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle programme. (Experimental): 8 month lifestyle programme.
  Interventions: Behavioral: 8-month group lifestyle programme

INTERVENTIONS:
Behavioral: 8-month group lifestyle programme — Dietary and lifestyle counselling (11 sessions), weekly exercise programme and 3 fasting blood samples at baseline, 4 and 8 months.

SUMMARY:
The aim of this study is to investigate weather gradual weight loss achieved with healthy lifestyle changes influence hormonal factors affecting appetite and blood glucose control in obese people without presence of diabetes.

DETAILED DESCRIPTION:
Obesity is becoming a growing and significant public health problem. Evidence from various national surveys over the last 25 years show that the prevalence of obesity and overweight in adults in England has increased threefold. There is still no clear evidence available to explain the epidemic levels of obesity. A number of neuro-endocrine factors have a role in the regulation of food intake and in the control of insulin secretion. We are particularly interested in measuring levels of a hormone called Glucagon-like peptide 1 (GLP-1) which is released from the intestine when food is absorbed. This hormone in turn has an influence on the production of insulin and another hormone, glucagons, both of which are involved in controlling blood glucose ('blood sugar') levels and appetite control.

There is some evidence, that obese people with normal blood sugar control show attenuated GLP-1 levels, however the evidence is contradictive and statistical significance is unclear. There is an ample of evidence that in established diabetes GLP-1 levels are attenuated, however it still remains uncertain whether the lower GLP-1 levels contribute to the pathogenesis of the condition or are a consequence of chronic hyperglycaemia or other hormonal and metabolic changes, though the observation that GLP-1 levels are lower in obese subjects suggests the possibility that the former may be the case.

Recently Bournemouth Diabetes and Emdocrine Centre (BDEC) conducted a research trial on effect of weight loss on GLP-1 levels in subjects with new onset type 2 diabetes. After 8 months intensive lifestyle programme average weight loss was 7.8 kg with significant and sustained improvements in clinical and metabolic parameters. Despite this, the GLP-1 levels remained unchanged.

None of the previous studies looked how gradual healthy lifestyle changes with sensible weight loss goals and increased activity levels effect GLP-1 levels in obese non-diabetic population.

ELIGIBILITY:
Inclusion criteria:

1. BMI between 30-39.9kg/m2
2. Family history of diabetes (self reported)
3. Normal and impaired glucose tolerance
4. Obtain informed consent

Exclusion criteria:

1. BMI less than 30kg/m2 or more than 39.9kg/m2
2. Presence of diabetes or any other chronic disease or disability that might interfere with the study results
3. Anti-obesity or any other prescription medications that may interfere with the study results
4. Pregnancy
5. Unable to converse competently in English as special arrangements would need to be made for such people and this would be impractical in a group setting
6. Attending another weight management programme
7. Patients who would be unable to attend at least 75% of the programme sessions for medical or other reasons
8. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To estimate the correlation between weight loss over 8 months achieved through a programme of intensive lifestyle management and changes in GLP-1 production over the same period in obese without presence of diabetes but with family history of diabetes. | 8 month lifestyle programme

SECONDARY OUTCOMES:
The secondary aim is to examine the changes in weight, cardiovascular risk factors and hormonal regulators of food intake and blood glucose metabolism. | 8 months lifestyle programme

CONTACTS AND LOCATIONS:
Overall Officials: Dr Joe Begley, Principal Investigator — The Royal Bournemouth Hospitals
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom